CLINICAL TRIAL: NCT04586504
Title: Dose-Finding Study of Intranasal Midazolam for Procedural Sedation in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Emergency Medicine Foundation (Other); Mailman School of Public Health (Unknown)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Professor of Pediatrics in Emergency Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAS7996
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Procedural Anxiety
Keywords: Intranasal; Midazolam; Pediatric; Laceration repair; Sedation; Anxiolysis; Adaptive trial design; Dose finding
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Sequential selection procedure
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0.2 mg/kg (Experimental): Children in a single urban pediatric emergency department (ED) randomized to receive IN midazolam at 0.2 mg/kg.
  Interventions: Drug: Intranasal midazolam
- 0.3 mg/kg (Experimental): Children in a single urban pediatric emergency department (ED) randomized to receive IN midazolam at 0.3 mg/kg.
  Interventions: Drug: Intranasal midazolam
- 0.4 mg/kg (Experimental): Children in a single urban pediatric emergency department (ED) randomized to receive IN midazolam at 0.4 mg/kg.
  Interventions: Drug: Intranasal midazolam
- 0.5 mg/kg (Experimental): Children in a single urban pediatric emergency department (ED) randomized to receive IN midazolam at 0.5 mg/kg.
  Interventions: Drug: Intranasal midazolam

INTERVENTIONS:
Drug: Intranasal midazolam — 5 mg/mL concentration of midazolam. Maximum dose = 10 mg. Administered using a mucosal atomization device.
  Other Names: IN midazolam

SUMMARY:
Dose-finding study to compare intranasal midazolam doses of 0.2, 0.3, 0.4 and 0.5 mg/kg in children undergoing laceration repair to achieve the following aims:

Specific Aim #1: To determine the most effective dose of intranasal midazolam for producing adequate sedation state associated with each dose.

Specific Aim #2: To determine the time to recovery and describe the adverse events associated with each dose.

DETAILED DESCRIPTION:
Intranasal midazolam is a common and effective sedative whose use in children presenting to emergency departments has been described. However, the doses of intranasal midazolam used have varied greatly, with no identified optimal dose. Doses most commonly described in literature reviews, research studies, and clinical guidelines range from 0.2 to 0.5 mg/kg. There is only one study, retrospective, that compares doses and suggests that clinical efficacy is improved with higher doses, without any clear difference in safety. There is a need for a rigorously-conducted trial to determine the dose of intranasal midazolam that optimizes the adequacy of sedation state without leading to adverse events or compromising emergency department-centric outcomes such as time to onset of sedation and time to recovery. To fill this important and persistent gap in knowledge, the investigator will conduct a dose-finding study using an adaptive trial design to compare intranasal midazolam doses of 0.2, 0.3, 0.4, and 0.5 mg/kg in children undergoing laceration repairs, one of the most common types of minor trauma treated in emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 months to 7 years old (i.e. before their 8th birthday)
* Simple laceration
* Attending physician has decided intranasal midazolam indicated to facilitate repair

Exclusion Criteria:

* Repair using tissue adhesive (e.g. Dermabond) or staples
* Known or confirmed developmental delay
* Baseline motor neurological abnormality (e.g. motor deficit, cerebral palsy)
* Autism spectrum disorder
* Illness associated with chronic pain
* Known allergy to midazolam or any other benzodiazepine
* Eyelid laceration
* Tongue or intraoral lacerations
* Nasal obstruction that cannot be easily cleared
* Does not speak English or Spanish
* Foster children, wards of the state

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- NewYork Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsze DS, Ieni M, Fenster DB, Babineau J, Kriger J, Levin B, Dayan PS. Optimal Volume of Administration of Intranasal Midazolam in Children: A Randomized Clinical Trial. Ann Emerg Med. 2017 May;69(5):600-609. doi: 10.1016/j.annemergmed.2016.08.450. Epub 2016 Nov 4. PMID 27823876
- [Background] Cravero JP, Askins N, Sriswasdi P, Tsze DS, Zurakowski D, Sinnott S. Validation of the Pediatric Sedation State Scale. Pediatrics. 2017 May;139(5):e20162897. doi: 10.1542/peds.2016-2897. PMID 28557732
- [Background] Mellion SA, Bourne D, Brou L, Brent A, Adelgais K, Galinkin J, Wathen J. Evaluating Clinical Effectiveness and Pharmacokinetic Profile of Atomized Intranasal Midazolam in Children Undergoing Laceration Repair. J Emerg Med. 2017 Sep;53(3):397-404. doi: 10.1016/j.jemermed.2017.05.029. PMID 28992870
- [Background] Leu C-S, Levin B. On the probability of correct selection in the Levin-Robbins sequential elimination procedure. Stat Sin 1999;9(3):879-91.
- [Background] Malviya S, Voepel-Lewis T, Tait AR, Merkel S, Tremper K, Naughton N. Depth of sedation in children undergoing computed tomography: validity and reliability of the University of Michigan Sedation Scale (UMSS). Br J Anaesth. 2002 Feb;88(2):241-5. doi: 10.1093/bja/88.2.241. PMID 11878656
- [Background] Bhatt M, Kennedy RM, Osmond MH, Krauss B, McAllister JD, Ansermino JM, Evered LM, Roback MG; Consensus Panel on Sedation Research of Pediatric Emergency Research Canada (PERC) and the Pediatric Emergency Care Applied Research Network (PECARN). Consensus-based recommendations for standardizing terminology and reporting adverse events for emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2009 Apr;53(4):426-435.e4. doi: 10.1016/j.annemergmed.2008.09.030. Epub 2008 Nov 20. PMID 19026467
- [Background] Elliott CH, Jay SM, Woody P. An observation scale for measuring children's distress during medical procedures. J Pediatr Psychol. 1987 Dec;12(4):543-51. doi: 10.1093/jpepsy/12.4.543. No abstract available. PMID 3430286
- [Result] Tsze DS, Woodward HA, McLaren SH, Leu CS, Venn AMR, Hu NY, Flores-Sanchez PL, Stefan BR, Shen ST, Ekladios MJ, Cravero JP, Dayan PS. Optimal Dose of Intranasal Midazolam for Procedural Sedation in Children: A Randomized Clinical Trial. JAMA Pediatr. 2025 Sep 1;179(9):979-986. doi: 10.1001/jamapediatrics.2025.2181. PMID 40720114

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
Started | 19 | 24 | 29 | 29
Completed | 19 | 24 | 29 | 29
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg | Total
Number analyzed (Participants) | 19 | 24 | 29 | 29 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 24 | 29 | 29 | 101
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2 [1 to 3] | 3 [2 to 3.8] | 4 [2.5 to 5] | 3 [2.5 to 5] | 3 [2 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 10 | 11 | 38
  Male | 13 | 13 | 19 | 18 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1 | 2
  Black | 2 | 0 | 2 | 4 | 8
  Hispanic | 13 | 17 | 24 | 21 | 75
  White | 2 | 7 | 1 | 3 | 13
  More than one race | 1 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 24 | 29 | 29 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Who Achieved PSSS Score 2, 3, or 4 for 95% or Greater of the Scored Procedure
Description: The Pediatric Sedation State Scale (PSSS) is scored from 0 to 5, representing a continuum of sedation that spans from over-sedation associated with changes in vital signs (0) to inadequate sedation (5).
Time Frame: From study drug administration until procedure finished (approximately 60 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
Number analyzed (Participants) | 19 | 24 | 29 | 29
Participants | 9 | 12 | 20 | 19

2. Secondary Outcome: Time to Recovery
Description: Time (in minutes) from procedure completion until a Simplified Aldrete Score (SAS) of at least 6 is achieved. The score ranges from 0 (lowest) to 8 (highest). If a patient already fulfills criteria for recovery at procedure start, then time to recovery is 0.
Time Frame: From study drug administration until patient discharge (approximately 120 minutes)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
Number analyzed (Participants) | 19 | 24 | 29 | 29
minutes | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Number of Adverse Events
Description: Adverse events will be defined using the Pediatric Emergency Research Canada and Pediatric Emergency Care Applied Research Network Consensus-Based Recommendations. These adverse events include oxygen desaturation; apnea (central, obstructive, laryngospasm); clinically apparent pulmonary aspiration; retching/vomiting; bradycardia; hypotension; excitatory movements; paradoxical response to sedation; unpleasant recovery reactions; and permanent complications (including death).
Time Frame: From study drug administration until patient discharge (approximately 120 minutes)
Measure: Number; unit: adverse events
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
Number analyzed (Participants) | 19 | 24 | 29 | 29
adverse events | 0 | 0 | 2 | 0

4. Secondary Outcome: Time to Onset of Minimal Sedation
Description: Time (in minutes) from administration of intranasal midazolam until a University of Michigan Sedation State (UMSS) score of 1 is achieved. The UMSS represents a spectrum of depth of sedation ranging from unarousable (4) to awake and alert (0). Note: This outcome was initially listed as a primary outcome, but was changed to a secondary outcome in the IRB-approved protocol and prior to enrollment of the first patient.
Time Frame: From study drug administration until procedure finished (approximately 60 minutes)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
Number analyzed (Participants) | 19 | 24 | 29 | 29
minutes | 4.2 [2.8 to 6.6] | 3.7 [3.1 to 5] | 3.9 [3.1 to 4.4] | 3.9 [3.3 to 5]

5. Secondary Outcome: UMSS Scale Score
Description: Depth of sedation will be measured using the University of Michigan Sedation Scale (UMSS). This sedation scale ranges from zero to four with higher numbers indicating deeper sedation.
Time Frame: From study drug administration until procedure finished (approximately 60 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
Number analyzed (Participants) | 19 | 24 | 29 | 29
Participants
  UMSS = 0 | 3 | 2 | 1 | 2
  UMSS = 1 | 16 | 22 | 28 | 27
  UMSS = 2, 3 or 4 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of intranasal midazolam administration until discharge from emergency department (approximately 120 minutes)
Arm/Group | 0.2 mg/kg | 0.3 mg/kg | 0.4 mg/kg | 0.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/24 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/24 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/19 | 0/24 | 2/29 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.2 mg/kg (N=19) | 0.3 mg/kg (N=24) | 0.4 mg/kg (N=29) | 0.5 mg/kg (N=29)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paradoxical reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT04586504/Prot_SAP_000.pdf